CLINICAL TRIAL: NCT06352320
Title: Risk Stratification and New Early Prevention and Treatment Strategies for Patients With Cardiomyopathy (STRENGTH Trial): a National Multi-center, Retrospective-prospective, Cohort Study
Brief Title: Risk Stratification and New Early Prevention and Treatment Strategies for Patients With Cardiomyopathy (STRENGTH）
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-533
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Cardiomyopathies
Keywords: Cardiomyopathies; Prognostic factors
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For the retrospectively enrolled patients, we will collect their biological samples previously housed in the Biobank of The First Affiliated Hospital of Xi'an Jiaotong University.
  For the prospectively enrolled patients, we will collect a variety of biological samples at admission, before discharge, 1st, 3rd, 6th, 9th month, 1st, 2nd, 3rd year after discharge, including blood, urine, feces, other types of body fluids (such as pericardial effusion), tissue samples from surgery and biopsy (such as pericardial effusion, myocardial tissue, tumors, blood clots, etc.), or samples that need to be disposed of as medical waste (blood clots, etc.), or the sample itself requires pathological examination to assist in diagnosis and treatment (e.g. endocardial muscle biopsy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HCM group: Patients were diagnosed with HCM.
  Interventions: Biological: Diagnosis of HCM
- DCM group: Patients were diagnosed with DCM.
  Interventions: Biological: Diagnosis of DCM
- ARVC group: Patients were diagnosed with ARVC.
  Interventions: Biological: Diagnosis of ARVC
- NDLVC group: Patients were diagnosed with NDLVC.
  Interventions: Biological: Diagnosis of NDLVC
- RCM group: Patients were diagnosed with RCM.
  Interventions: Biological: Diagnosis of RCM
- LVNC group: Patients were diagnosed with LNVC.
  Interventions: Biological: Diagnosis of LVNC

INTERVENTIONS:
Biological: Diagnosis of HCM — Hypertrophic cardiomyopathy (HCM) is defined as the presence of increased LV wall thickness (with or without RV hypertrophy) or mass that is not solely explained by abnormal loading conditions.
  Groups: HCM group
Biological: Diagnosis of DCM — Dilated cardiomyopathy (DCM) is defined as the presence of LV dilatation and global or regional systolic dysfunction unexplained solely by abnormal loading conditions (e.g. hypertension, valve disease, CHD) or CAD.Very rarely, LV dilatation can occur with normal ejection fraction (EF) in the absence of athletic remodelling or other environmental factors; this is not in itself a cardiomyopathy, but may represent an early manifestation of DCM. The preferred term for this is isolated left ventricular dilatation. Right ventricular dilatation and dysfunction may be present but are not necessary for the diagnosis.
  Groups: DCM group
Biological: Diagnosis of ARVC — Arrhythmogenic right ventricular cardiomyopathy (ARVC) is defined as the presence of predominantly RV dilatation and/or dysfunction in the presence of histological involvement and/or electrocardiographic abnormalities in accordance with published criteria.
  Groups: ARVC group
Biological: Diagnosis of NDLVC — The NDLVC phenotype is defined as the presence of non-ischaemic LV scarring or fatty replacement regardless of the presence of global or regional wall motion abnormalities (RWMAs), or isolated global LV hypokinesia without scarring.
  Groups: NDLVC group
Biological: Diagnosis of RCM — Restrictive cardiomyopathy (RCM) is defined as restrictive left and/or RV pathophysiology in the presence of normal or reduced diastolic volumes (of one or both ventricles), normal or reduced systolic volumes, and normal ventricular wall thickness.Restrictive cardiomyopathy commonly presents as biatrial enlargement. Left ventricular systolic function can be preserved, but it is rare for contractility to be completely normal. Restrictive pathophysiology may not be present throughout the natural history, but only at an initial stage (with an evolution towards a hypokinetic-dilated phase). Restrictive physiology can also occur in patients with end-stage hypertrophic and dilated cardiomyopathy; the preferred terms are 'hypertrophic' or 'dilated cardiomyopathy with restrictive physiology'. Restrictive ventricular physiology can also be caused by endocardial pathology (fibrosis, fibroelastosis, and thrombosis) that impairs diastolic function
  Groups: RCM group
Biological: Diagnosis of LVNC — The term 'left ventricular non-compaction' (LVNC) has been used to describe a ventricular phenotype characterized by prominent LV trabeculae and deep intertrabecular recesses. The myocardial wall is often thickened with a thin,compacted epicardial layer and a thickerendocardial layer. Left ventricular non-compaction is frequently a familial trait and is associated with variants in a range of genes, including those encoding proteins of the sarcomere, Z-disc, cytoskeleton, and nuclear envelope. Left ventricular non-compaction has also been used to describe an acquired and sometimes transient phenomenon of excessive LV trabeculation (e.g. in athletes, during pregnancy, or following vigorous activity)that must reflect increased prominence of an otherwise normal myocardial architecture, given that cardiomyocytes are terminally differentiated and the formation of new cardiac structures is impossible.The Task Force does not consider LVNC to be a cardiomyopathy in the general sense.
  Groups: LVNC group

SUMMARY:
This study will include patients with different types of cardiomyopathy from multiple centers were prospectively enrolled in a retrospective study to establish a natural population cohort of cardiomyopathy patients. By collecting clinical data and biological samples from surgical patients, we will construct a prognostic system for cardiomyopathy, optimize risk stratification, explore new strategies for the early prevention and treatment of cardiomyopathy, and improve the efficiency of clinical cardiomyopathy patients' diagnosis and treatment.

DETAILED DESCRIPTION:
This study will include patients with different types of cardiomyopathy from multiple centers were prospectively enrolled in a retrospective study to establish a natural population cohort of cardiomyopathy patients. By collecting clinical data and biological samples from surgical patients, we will construct a prognostic system for cardiomyopathy, optimize risk stratification, explore new strategies for the early prevention and treatment of cardiomyopathy, and improve the efficiency of clinical cardiomyopathy patients' diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* The diagnosis of cardiomyopathy was confirmed by cardiac ultrasound, electrocardiogram, magnetic resonance angiography, pathological examination and gene sequencing.
* Patients or their families agreed to participate in the study and authorized informed consent.

Exclusion Criteria:

* Incomplete clinical data.
* Do not agree to the inclusion or refuse to authorize the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cardiomyopathy at all centers including The First Affiliated Hospital of Xi'an Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of mortality rate | At diagnosis, before discharge (about 7 days), 1, 3, 6, 9 month, 1, 2, 3, 5, 10 year.
  The survival status will be obtained from the medical records and phone calls to patients or their family members

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China